CLINICAL TRIAL: NCT05813080
Title: Computer-assisted Risk Evaluation in the Early Detection of Psychotic Disorders
Acronym: CARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HeinrichHeine
Record Dates: First submitted 2023-03-14; First posted 2023-04-14 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Psychotic Disorders; Prevention
Keywords: Psychosis-Risk Syndromes; high-risk; Cognitive Disturbances; Artificial Intelligence
MeSH Terms: conditions — Psychotic Disorders; Cognition Disorders

STUDY DESIGN:
Intervention Model Description: The aim of risk-adapted treatment (RAB) arm is to reduce the number of patients with an increased clinical risk for psychosis to actually develop a manifest psychosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARE interventional treatment (Experimental): AI-computerassisted prognosis of high risk psychosis profile and adapted study-specific therapy taking place in early-recognition centers.
  Interventions: Device: "pronia.ai" medical device for high risk psychosis prognosis
- Standard of Care Control arm (Active Comparator): Treatment as usual (TAU) patient will receive their usual treatment from their local physicians and therapeutic personnel.
  Interventions: Other: Treatment-as-usual (TAU)

INTERVENTIONS:
Device: "pronia.ai" medical device for high risk psychosis prognosis — In addition to the computer-assisted prognosis of risk for reaching a psychosis, all patients assigned to the active treatment arm will receive additional in-depth clinical diagnostics including neuropsychological testing. Adapted psychological treatment will be offered consisting of 16 to 24 sessions over a period of six months.
  Arms: CARE interventional treatment
Other: Treatment-as-usual (TAU) — Referral back to the previous care system. Further treatment is left to the referring primary care providers.
  Arms: Standard of Care Control arm

SUMMARY:
Multicenter randomized controlled trial (RCT) with artificial intelligence (AI)-staged early diagnostics and risk-adapted treatment (RAB) as interventional treatment arm and treatment-as-usual (TAU) as control treatment arm for patients with an increased clinical risk for psychosis.

DETAILED DESCRIPTION:
The study is a Investigator Initiated Trial (IIT)/Other clinical trial of a class 2a medical device according to article 82 medical devices regulation of the European Union.

The aim of risk-adapted treatment (RAB) arm is to reduce the number of patients with an increased clinical risk for psychosis to actually develop a manifest psychosis.

Patients assigned to the active treatment arm will receive additional in-depth clinical diagnostics including neuropsychological testing.

The AI-supported algorithm "pronia.ai" uses information from both the individual patient data of the specialized routine diagnostics as well as from in-depth clinical diagnostics.

There are two predictions, an individual quantitative assessment of the individual risk of transition to psychosis and the individual prognosis with regard to the level of psychosocial functioning 12 months after inclusion in the study.

The therapists and patients receive a non-binding risk profile from the AI-based recommendation to adjust the treatment intensity from 16 to 24 sessions over a period of six months.

The cognitive behavioral therapy-based manual "Integrated Preventive Psychological Preventive Psychological Intervention (IPPI)" manual is used. In the treatment-as-usual arm (TAU),the patients receive referral back to the previous care system; further treatment (and additional diagnostics, if necessary) is left to the referring primary care providers.

ELIGIBILITY:
Inclusion Criteria:

* The increased risk of psychosis includes either a symptomatic "ultra high-risk" stage of the Structured Interview for Psychosis-Risk Syndromes or the "Cognitive Disturbances" risk criterion of the Schizophrenia Proneness Instrument - Children and Youth and Adult versions
* ages 16 to 40
* Presence of a written informed consent from the patient and, if applicable, the legal guardian.

Exclusion Criteria:

* manifest psychosis according to the definition of the Structured Interview for Psychosis-Risk Syndromes (according to the PRONIA-study) (At least one P-syndrome with a rating of 6 on a daily frequency and for a period of more than one week)
* Lack of capacity to give consent (the patient lacks the capacity to consent if the individual case with regard to the specific treatment measure is excluded. Only when the physician has concrete indications that the patient's capacity to consent may be lacking, he may and must must examine it. Mental disorders (e.g. delirium, dementia, psychosis, mania, depression) or cognitive impairments can have an influence on the capacity to consent. Indications for doubts of a ability to give informed consent exist if the physician has the impression that the patient is not able to understand the provided patient information and is not able to reproduce essential information about the study in his or her own words and is not aware of the possible consequences of the proposed measures
* Severe suicidality during the recruitment phase (CDSS items 8 ≥2)
* A current or past neurological disease of the brain.
* a current or past known somatic disease that potentially affects the structure or function of the brain
* Antipsychotic medication in the indication treatment of psychotic symptoms for >30 days (cumulative number of days) at or above the starting dose for psychosis according to the current German Association for Psychiatry, Psychotherapy and Psychosomatics (DGPPN) S3 guidelines.
* an antipsychotic medication in the indication treatment of psychotic symptoms in the 3 months prior to the initial examination (regardless of the duration of use) at or above the starting dose for psychosis according to the current DGPPN S3 guidelines
* An inadequate level of hearing for neurocognitive testing
* a current or past head trauma with unconsciousness (>5 min).
* a current or past alcohol dependence (ICD-10 F10.x)
* A current polytoxicomania (multiple substance dependence) or polytoxicomania in the past 6 months (ICD-10 F19.x)
* Presence of medical reasons that contraindicate performance of an MRI
* Insufficient language skills to understand the indication and the purpose of the intended examinations and interventions
* stationary accommodation against the patient's will

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 260 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Structured Interview for Psychosis-Risk Syndromes (SIPS) | 12-month after inclusion
  Presence of psychotic syndrome (POPS) criteria as modified according to the "PRONIA" study, resulting in a score of 0= "no psychosis" or 1= "psychosis"

SECONDARY OUTCOMES:
Internalized Stigma of Mental Illness Scale (ISMI) | 12-month after inclusion
  Consisting of 5-subscales, comprising of 29 items in total using response formats varying from 4-point Likert scales (1='not at all', 4='very often') to 5-point Likert scales (1='never', 5='very often'), assessing self-stigma in terms of alienation, adoption of stereotypes, experiences of discrimination, social withdrawal and stigma resistance.
Stigma-Stress-Scale | 12-month after inclusion
  two dimensions are assessed, 8 items are rated on a 5-point Likert-scale from "strongly disagree" to "totally agree", capturing self-assessed-stigma stress.
Self-Identification of Mental Illness Scale (SELF-I) | 12-month after inclusion
  5-point Likert-scale ranging from 1 = "not true at all" to 5 = " is completely true", capturing the degree of self-identification with mental illnesses.
Coming-Out with Mental Illness Scale (COMIS) | 12-month after inclusion
  consisting of two subscales with 7 and 14 items, each with 7-step Likert-scale ranging from 1 = "do not agree at all" to 7 = " totally agree", capturing a potential change of strategies for dealing with mental illness.
Secrecy and disclosure-related distress - scale | 12-month after inclusion
  7-point single-item-scale ranging from 1 = " not at all" to 7 = "very much", measuring the degree of subjective stress.
Psychosis own health-concern single score | 12-month after inclusion
  5-point Likert-scale ranging from 1 = "not at all" to 5 = "strong", capturing the degree of self-concern in terms of getting a psychosis one day.
Numeracy Scale | 12-month after inclusion
  A single score from 0 to 100% indicating the patient self-estimated amount of belief in risk for developing psychosis within the next 12 months.
Coping (Ten-Flex) | 12-month after inclusion
  Patient self-estimation of likelihood for developing psychosis given on a visual analogue scale (VAS) indicating "I will not develop psychosis in the next 12 months" on the left side of the scale up to "I will definitely develop psychosis in the next 12 months" on the right side of the scale.
Risk Perception Scale | 12-month after inclusion
  A score from 1 =no risk" to 7 = "absolutely certain" indicating the risk for developing psychosis.
Risk Recall Scale | 12-month after inclusion
  A score from 1 = "much lower" to 5 "much higher" indicating the risk for developing psychosis compared to a healthy peer.
Health-related quality of life (EQ-5D) | 12-month after inclusion
  patient questionnaire consisting of two sub-scores. a) score from 0-10 whereas a higher score indicates greater impairment; b) score from 0-100 whereas a higher score indicates better current health status to measure the quality of Life.
Brief Multidimensional Life Satisfaction Scale (BMLSS) | 12-month after inclusion
  Score from 0-126, a higher score indicates a higher amount of satisfaction.
Client Sociodemographic and Service Receipt Inventory (CSSRI-EU) | 12-month after inclusion
  Changes in service use are measured with a semi-structured interview to assess social and demographic data, accommodation data, detailed information regarding treatment, professional visits and social and health service utilization for estimating healthcare costs. Additionally, the CSSRI systematically records the use of psychiatric, medical, psycho-social and rehabilitative health services (direct costs) and productivity losses (indirect costs) and therefore completely covers the costs of the disease from an economic perspective.
Patient Satisfaction Questionnaire (ZUF-8) | 12-month after inclusion
  8 Items with a total score of 8-32, ranging from 4 = "very satisfied" to 1="fairly satisfied" whereas a higher score indicates higher patient satisfaction.
Social and occupational assessment scale SOFAS | 12-month after inclusion
  Scores from 0-100, a higher score indicates better social functioning.
Global Functioning Social Scale (GF:S) | 12-month after inclusion
  Scores from 1-10, a higher score indicates better global functioning
Global Functioning Role Scale (GF:R) | 12-month after inclusion
  Scores from 1-10, a higher score indicates better functioning
Secrecy-Symptoms Scale | 12-month after inclusion
  Five questions (either yes or no) asking who the patient has told about the risk for developing psychosis

CONTACTS AND LOCATIONS:
Overall Officials: Eva Meisenzahl-Lechner, Prof., Principal Investigator — Klinik und Poliklinik für Psychiatrie und Psychotherapie LVR-Klinikum Düsseldorf
Locations (21):
- Germany (21):
  - ZfP Reichenau - Akademisches Lehrkrankenhaus Universität Konstanz, Konstanz, Baden-Wurttemberg
  - Zentralinstitut für Seelische Gesundheit, Mannheim, Baden-Wurttemberg
  - Klinik für Psychiatrie und Psychotherapie Universität Tübingen, Tübingen, Baden-Wurttemberg
  - Bezirkskrankenhaus Augsburg, Klinik für Psychiatrie, Psychotherapie und Psychosomatik der Universität Augsburg, Augsburg, Bavaria
  - Klinikum der Ludwig-Maximilians-Universität München, München, Bavaria
  - Zentrum für psychische Gesundheit, U11iversitätsklinikum Würzburg, Würzburg, Bavaria
  - Klinik für Psychiatrie, Psychotherapie und Psychosomatik, Universitätsklinikum Aachen, RWTH Universität Aachen, Aachen, North Rhine-Westphalia
  - LWL-Universitätsklinikum Bochum der Ruhr--Universität Bochum, Klinik für Psychiatrie, Psychotherapie und Präventivmedizin, Bochum, North Rhine-Westphalia
  - KJPP LVR-Klinik Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Bonn Klinik für Psychiatrie und Psychotherapie, Bonn, North Rhine-Westphalia
  - Uniklinik Köln, Klinik und Poliklin-ik für Psychiatrie, Psychosomatik und Psychotherapie des Kindes- und Jugendalters, Cologne, North Rhine-Westphalia
  - Klinik und Poliklinik für Psychiatrie und Psychotherapie Heinrich-Heine-Universität Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Institut für Translationale Psychiatrie, Münster, North Rhine-Westphalia
  - Rheinhessen Fachklinik Alzey, Alzey, Rhineland-Palatinate
  - UKD Dresden, Klinik und Poliklinik für Psychiatrie und Psychotherapie, Dresden, Saxony
  - Otto-von-Guericke- Universität Magdeburg, Magdeburg, Saxony-Anhalt
  - Zentrum für Integrative Psychiatrie Kiel, Kiel, Schleswig-Holstein
  - Zentrum für Integrative Psychiatrie (ZIP) und Fachklinik für Junges Leben (JuLe) Kinder- und Jugendpsychiatrie, Lübeck, Schleswig-Holstein
  - Vivantes Klinikum Am Urban, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinik und Poliklinik für Psychiatrie und Psychotherapie, Universitätsklinikum Hamburg-Eppendorf {UKE), Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bommhardt T, Peschl J, Schultze-Lutter F, Koutsouleris N, Meisenzahl E, Koberlein-Neu J; CARE Study Group. Enhancing early detection and treatment of psychosis in Germany: a protocol for the health economic evaluation of an artificial intelligence-guided complex intervention. BMJ Open. 2025 Jun 18;15(6):e103151. doi: 10.1136/bmjopen-2025-103151. PMID 40533222